CLINICAL TRIAL: NCT00351312
Title: Evaluation of Foot Pressure in Volunteers Wearing Socks Weaved With Pressure Reducing Soles
Brief Title: Creation of a Pressure Reducing Areas in Socks
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SHEBA-06-4163-UG-CTIL
Record Dates: First submitted 2006-07-11; First posted 2006-07-12 (Estimated); Last update posted 2006-07-12 (Estimated); Status verified 2006-07

CONDITIONS: Pressure Ulcers
Keywords: Pressure ulcers; socks; foot pressure
MeSH Terms: conditions — Pressure Ulcer

INTERVENTIONS:
Device: special socks

SUMMARY:
Evaluation of the ability of socks weaved with pressure relieving areas to reduce the pressure on the foot when weight bearing.

DETAILED DESCRIPTION:
Increased pressure in weight bearing areas of the foot, especially in insensate feet may lead to the development of pressure sore. The creation of socks with pressure relieving areas by special weaving technique may prevent the development of these complications.

Three (3) volunteers will be examined walking on a Tekscan pressure mat, barefoot and then wearing socks weaved in a new technique, from cotton, nylon and acrilan.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers

Exclusion Criteria:

* foot deformity

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4
Dates: Start 2006-06; Study Completion 2006-06

PRIMARY OUTCOMES:
Pressure measurement

CONTACTS AND LOCATIONS:
Overall Officials: Uri Givon, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Motion Analysis Laboratory, Sheba Medical Center, Tel Litwinsky, Israel